CLINICAL TRIAL: NCT07345195
Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen and MSM on Facial Erythema and Other Skin Parameters: Double Blind, Placebo-controlled, Randomised Three-way Study Comparing the Efficacy of Two Test Products
Brief Title: The Effect of 16-week Dietary Intake of Food Supplements Containing Collagen and MSM on Facial Erythema and Other Skin Parameters
Acronym: TO-COSKIN4
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VIST - Faculty of Applied Sciences (Other)
Collaborators: Tosla d.o.o. (Industry); Slovenian Research Agency (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIST TO-COSKIN4 12-2025
Record Dates: First submitted 2025-12-24; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Erythema; Telangiectasis; Skin Redness
Keywords: Facial telangiectasiae; Erythema; Facial erythema; Collagen; MSM; Dietary supplement; Skin health; Skin redness; Erythema-prone skin
MeSH Terms: conditions — Erythema; Telangiectasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IP1 group (Active Comparator): Participants will receive investigational product 1 containing collagen (10 g/ 30 mL), MSM (2.0 g/ 30 mL) and vitamin C (160 mg/ 30 mL) for 16 weeks.
  Interventions: Dietary Supplement: CPMSM-HD
- IP2 group (Active Comparator): Participants will receive investigational product 2 containing collagen (5 g/ 30 mL), MSM (1.5 g/ 30 mL) and vitamin C (160 mg/ 30 mL) for 16 weeks.
  Interventions: Dietary Supplement: CPMSM-LD
- Placebo group (Placebo Comparator): Placebo group participants will receive placebo syrup without active ingredients (0 mg of collagen, 0 mg of MSM and 0 mg of vitamin C), 30 mL/daily for 16 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: CPMSM-HD — Participants will test continuous administration of investigational product for 16 weeks.
  Other Names: Investigational product 1
  Arms: IP1 group
Dietary Supplement: CPMSM-LD — Participants will test continuous administration of the investigational product for 16 weeks.
  Other Names: Investigational product 2
  Arms: IP2 group
Dietary Supplement: Placebo — Participants will test continuous administration of placebo product for 16 weeks.
  Arms: Placebo group

SUMMARY:
The aim of this study is to compare the effects of 16 weeks of daily dietary supplementation with two investigational products containing collagen, methylsulfonylmethane (MSM), and vitamin C on skin parameters in comparison to a placebo product. The study will be conducted in healthy human subjects with visible facial erythema and telangiectasiae (cheeks), stable for ≥3 months, without active rosacea.

The primary objective is to demonstrate beneficial effects of the investigational products on facial erythema.

The secondary objective is to evaluate the effect of the investigational products on facial telangiectasiae severity.

Other skin parameters will be assessed as supportive endpoints, and differences in efficacy between the two investigational formulations will also be evaluated.

DETAILED DESCRIPTION:
This is a single-centre, randomized, double-blind, placebo-controlled, one-period effectiveness study designed to evaluate the effects of multiple-dose, daily dietary supplementation over a 16-week period on skin parameters in healthy human subjects. The study population consists of subjects with visible facial erythema and telangiectasiae predominantly on the cheeks, stable for at least 3 months prior to inclusion, and without clinical signs of active rosacea.

Eligible participants will be randomized to receive one of two investigational products or a placebo product, administered as a daily oral dose of 30 mL for 16 consecutive weeks. The investigational products contain the following compositions: Investigational Product 1 (IP1): collagen 10 g, methylsulfonylmethane (MSM) 2.0 g, and vitamin C 160 mg; and Investigational Product 2 (IP2): collagen 5 g, MSM 1.5 g, and vitamin C 160 mg.

The primary objective of the study is to evaluate whether 16 weeks of supplementation with the investigational products results in a beneficial effect on facial erythema compared with placebo. The secondary objective is to assess the effect of the investigational products on facial telangiectasiae severity.

Supportive objectives include the evaluation of additional skin parameters and the assessment of differences in efficacy between the two investigational formulations.

ELIGIBILITY:
Inclusion criteria:

* Caucasian female volunteers aged 35 to 65 years at the time of signing the Informed Consent Form (ICF).
* Signed Informed Consent Form (ICF).
* Fitzpatrick skin phototypes I-IV.
* Presence of visible signs of skin ageing.
* Presence of visible facial telangiectasias, primarily on the cheeks.
* Presence of facial erythema with a baseline score ≤ 3 on the 5-point Clinical Erythema Assessment (CEA) scale.
* Stable erythema-prone facial skin for at least 3 months prior to study inclusion, without clinical signs of active rosacea.
* In good general health, as determined by medical history.
* Body Mass Index (BMI) < 35.
* Willingness and ability to:

  * Comply with all study procedures and complete a subject diary.
  * Maintain usual lifestyle habits throughout the study.
  * Not initiate or modify oestrogen or progesterone therapies during the study.
  * Maintain the same cosmetic and skincare routine and comply with sun protection guidelines throughout the study.
  * Avoid rejuvenation treatments during the study.
  * Refrain from consuming food supplements containing collagen or other protein-based supplements, methylsulfonylmethane (MSM), or anti-inflammatory and/or antioxidant compounds with a known or potential impact on skin inflammation or vascular response for the duration of the study.

Exclusion criteria:

* Pregnancy or breastfeeding.
* Vegan diet.
* Heavy smoking or frequent alcohol-induced flushing.
* Occupational or hobby-related excessive heat exposure (e.g. chefs, sauna workers) likely to interfere with vascular stability.
* Anticipated sunbathing or solarium use, or major planned changes in sun exposure before or during the study.
* Planned major changes during the study in:

  * Skincare routine
  * Hormonal therapy (contraception or hormone replacement therapy)
* Significant changes in dietary habits or dietary supplementation within 3 months prior to inclusion.
* Regular use within 3 months prior to inclusion of food supplements containing:

  * Methylsulfonylmethane (MSM);
  * Collagen or other protein-based supplements;
  * Anti-inflammatory supplements (e.g. bioflavonoids/rutin, curcumin, EPA) and/or antioxidant supplements with a known or potential impact on skin inflammation or vascular response.
* Any diagnosed, uncontrolled, untreated, or unstable medical condition.
* Clinically significant history of metabolic, gastrointestinal, hepatic, renal, or haematological disease.
* Mental incapacity or psychiatric condition that may impair understanding of the study or compliance with study requirements.
* Any clinically significant acute or chronic inflammatory skin disease, including but not limited to acne, perioral dermatitis, psoriasis, atopic dermatitis, or lupus.
* Skin pigmentation disorders at the assessment sites.
* Active rosacea within 3 months prior to study entry, defined as the presence of papules/pustules, frequent flushing episodes typical of rosacea, or ocular involvement.
* Frequent vasomotor hot flushes (e.g. perimenopausal or menopausal), which may interfere with erythema assessments.
* Use of medications affecting skin or vascular reactivity, including but not limited to: systemic corticosteroids, anticoagulants (e.g. coumarins, heparin), vasodilators (e.g. hydralazine, nitroglycerin), antibiotics with potential to affect erythema or vascular response, immunomodulators, regular or long-term use of non-steroidal anti-inflammatory drugs (NSAIDs)
* Use of systemic retinoids within 3 months prior to study entry.
* Changes of skin care routine regimen within 4 weeks prior to study entry.
* Use of highly concentrated topical products (>15% azelaic acid, 10% vitamin C…) affecting inflammatory or vascular facial responses within 4 weeks prior to study entry.
* Invasive rejuvenation treatments (e.g. medium or deep chemical peels, ablative or vascular laser therapies) within 6 months prior to study entry.
* Non-invasive or minimally invasive rejuvenation treatments (e.g. microneedling, mesotherapy, superficial chemical peels, radiofrequency, electrotherapy, ultrasound, IPL) within 3 months prior to study entry.
* Known or suspected allergy to any ingredient of the investigational product(s).

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 90 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change of redness score from baseline in test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational products on redness score after 16 weeks of dietary supplementation will be assessed using Antera 3D CS, as a 0-100 score. Differences between test groups will also be evaluated.
Change of redness variation from baseline in test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational products on redness variation after 16 weeks of dietary supplementation will be assessed using Antera 3D CS in arbitrary units (a.u.).
Change of hemoglobin hyperconcentration area from baseline in test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational products on the hemoglobin hyperconcentration area after 16 weeks of dietary supplementation will be assessed using Antera 3D CS in mm². Differences between test groups will also be evaluated.
Change of hemoglobin hyperconcentration intensity from baseline in test groups in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  Assessment of the effects of the investigational products on the hemoglobin hyperconcentration intensity after 16 weeks of dietary supplementation will be assessed using Antera 3D CS in arbitrary units (a.u.).

SECONDARY OUTCOMES:
Change of visibility of facial telenagiectasiae from baseline in test groups, in comparison to placebo group after 16 weeks of dietary supplementation | 16 weeks
  The effects of the investigational product on facial telangiectasia after 16 weeks of dietary supplementation will be assessed using expert evaluation using Telangiectasia in Rosacea Severity Assessment (TRoSA) scale on a 0-4 grade (0 - No visible telangiectasia, 4 - Extensive, dense, and highly visible telangiectasia involving a large surface area).

CONTACTS AND LOCATIONS:
Overall Officials: Katja Žmitek, PhD, Study Director — Head of Reasearch Group
Locations (1):
- VIST - Faculty of Applied Sciences, Institute of Cosmetics, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No